CLINICAL TRIAL: NCT03741764
Title: Treatment of Dupuytren's Disease With Minimal Invasive Surgery and VIVOSORB® Resorbable Implant Device
Acronym: Vivosorb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: prof. dr. Ilse Degreef (Other)
Responsible Party: Sponsor-Investigator, prof. dr. Ilse Degreef, Prof. Dr. Ilse Degreef, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S61390
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Dupuytren Contracture; Dupuytren Disease of Palm and Finger
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vivosorb (Other): Only arm in study
  Interventions: Device: Vivosorb

INTERVENTIONS:
Device: Vivosorb — Resorbable implant device

SUMMARY:
Dupuytren's disease is a progressive fibroproliferative condition of the hand which progresses in 20% of patients into a serious condition. In Flanders, Dupuytren's disease was found to be present in 32% of the population over 50 years.

In severe flexion contracture finger deformity due to Dupuytren's disease, functional loss of the finger (often the fourth or fifth digit) is significant.

Surgery remains the most efficient treatment for the correction of flexion deformities. Minimal invasive surgery with the creation of firebreaks for the fibrous strands causing this disease, withholds fast recovery. However, recurrence after surgery is not rare with numbers varying from 30 to 70% depending on fibrosis diathesis score of Abe, severity of the deformation and follow-up period.

Numerous surgical techniques have been used for Dupuytren disease, ranging from minimally invasive surgery to subtotal preaxial amputation with skin grafting.3 In this study a well-known technique faciectomie will be performed. During this surgery a device will be inserted called VIVOSORB® VIVOSORB® is a flexible bioresorbable polymer film which is designed to separate opposing tissues throughout the critical healing process. It is very flexible facilitating the surgeon to optimally position the sheet during surgery. It is made of 100% synthetic bioresorbable material and can be used in a variety of soft tissue surgery applications. VIVOSORB® provides a barrier function enabling the tissue to regenerate without interconnective attachment.

In the past cellulose, a biologic inert implant, was used for augmenting the effect of the surgical firebreaks . Cellulose has been proven to improve outcome. Nowadays, cellulose is not available for use during faciectomie surgery, since medical production has been ceased. VIVOSORB® can be a valid alternative.

DETAILED DESCRIPTION:
* Trial objectives The objective of this study is to establish if this device is a viable option for treating finger deformity caused by Dupuytren's disease. The main goal is to evaluate the efficacy and performance of this flexible bioresorbable polymer film (VIVOSORB®) Expected outcome is significant correction of the finger extension lack with preserved active finger flexion, without amputation risk or neurovascular damage due to more invasive surgery.
* Primary endpoints The device will be considered efficient if the pre-operative lack of finger extension (TPED) compared to the extension at two years post-operative improves by 46°.
* Secondary endpoints

Patient scores will be evaluated:

* Dash score
* EQ-5D-3L
* VAS pain & satisfaction Amputation is a final endpoint for this study. Secondary a comparison will be made between the population of this study and the population of a previous study in this center³ . In concrete terms this means that the improvement in finger extension will be compared between the VIVOSORB® group, the control³ and the cellulose group³.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with the disease of Dupuytren
* Subject suffers from a severe flexion deformity of the finger(s)
* Stage of Dupuytren's disease ≥ 3 as introduced by Tubiana4
* Dupuytren's patients with risk score D of Abe > 4 [5]
* Subject is 18 years or older
* Subject is willing to sign and date an IRB/EC-approved consent form
* Subject receives treatment in UZ Leuven

Exclusion Criteria:

* Subject is younger than 18
* Subject is not a good candidate for the study based on Investigator opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Total Passive Extension Deficit (TPED) | 2 years post-surgery
  TPED of the metacarpophalangeal, proximal interphalangeal and distal interphalangeal joints of each finger will be measured with an goniometer by an orthopaedic surgeon (the active and passive range of motion flexion and extension).

SECONDARY OUTCOMES:
DASH score | 2 years post-surgery
  This questionnaire asks the patient about their symptoms as well as their ability to perform certain activities. It's a 30 item questionnaire scored on a Likert scale from 1 (best outcome) to 5 (worst outcome). Maximum total DASH score=100. Higher DASH score indicates worse situation.
VAS pain & satisfaction | 2 years post-surgery
  On a 10 point scale the patients will score the pain of the hand and the level of satisfaction with the current state of their finger. 0=no pain, 10=worst pain; 0=not satisfied, 10=very satisfied
EQ-5D-3L | 2 years post-surgery
  Standardised instrument for use as a measure of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: No